CLINICAL TRIAL: NCT03714347
Title: The Effect of Cerebral Oxygenation on Postoperative Recovery in Intracranial Surgery
Acronym: Oxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Clinical Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TÜTF-BAEK 2016/225; TÜTF-BAEK (Registry Identifier: Local Ethic)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Intracranial Neoplasm
Keywords: cerebral oxygen monitoring; intracranial surgery; general anesthesia
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Control (Active Comparator): routine monitoring will be applied to this group
  Interventions: Device: routine monitoring
- Group Oxygen (Active Comparator): cerebral oxygen monitoring is applied to this group
  Interventions: Device: cerebral oxygen monitoring

INTERVENTIONS:
Device: cerebral oxygen monitoring — probes will be placed on eyebrows on forehead
  Arms: Group Oxygen
Device: routine monitoring — We will use routine monitoring intervention such as hate rate, arterial pressure, BIS. cerebral oxygen monitoring will not be applied to this group
  Arms: Group Control

SUMMARY:
The aim of this study was to investigate the effect of cerebral oxygenation on postoperative compilation in intracranial surgery.

DETAILED DESCRIPTION:
Patients undergoing intracranial surgery will be divided into two groups; group (Group Control n = 100) and cerebral oxygenation monitoring group (Group Oxygen). all hemodynamic parameters such as systolic blood pressure and diastolic blood pressure, oxygen saturation, Et CO2, SpO2;% and BIS during anesthesia during anesthesia will be recorded intraoperatively and 10 postoperatively in 5 min intervals. After extubation, Modified Aldrete Score, GKS (Glasgow Coma Scale), Ramsey Sedation Scale (RSS), nausea-vomiting and pain will be recorded in the recovery room. Pain assessment will be done with Visual Analog Scale (VAS). Patient satisfaction will be recorded. MMST (mini mental state test) and ASEM (antisaccadic eye movement test) tests will be performed preoperatively and postoperatively at 1st, 2nd and 3rd days.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial surgery will be performed
* Age 25-75
* ASA in the I-II-III risk group

Exclusion Criteria:

* Under GKS 15
* heart failure,
* renal insufficiency,
* liver failure,
* congenital neurological deficits

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12-28 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
cerebral oxygen monitoring data | cerebral oxygen values reported will be measured at 10 min intervals (intraoperative) and It would be reported by the first postoperative 10 minute intervals up to 30 minutes
  cerebral oxygen monitoring will measure peroperative

CONTACTS AND LOCATIONS:
Overall Officials: Emre Deren, MD, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Centrum, Turkey (Türkiye)